CLINICAL TRIAL: NCT01156311
Title: An Open-Label, Multicenter Study in Subjects With Relapsing-Remitting Multiple Sclerosis to Evaluate the Safety of 240 mg BG00012 TID Administered as Add-On Therapy to Beta Interferons (IFNβ) or Glatiramer Acetate (GA)
Brief Title: BG00012 Phase 2 Combination Study in Participants With Multiple Sclerosis
Acronym: EXPLORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109MS201
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis
Keywords: BG00012; MS; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glatiramer acetate (GA) and dimethyl fumarate (Experimental): Participants taking a stable dose of GA for at least 12 months prior to the study remain on that dose throughout the study. Dimethyl fumarate is administered at 120 mg three times a day (TID) on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
  Interventions: Drug: dimethyl fumarate
- Interferon beta (IFNβ) and dimethyl fumarate (Experimental): Participants taking a stable dose of one of the IFNβ products for at least 12 months prior to the study remain on that product and dose throughout the study. Dimethyl fumarate is administered at 120 mg three times a day (TID) on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — Days 1-7: 120 mg three times a day (TID) for a total daily dose of 360 mg. Day 8 to Week 24: 240 mg TID for a total daily dose of 720 mg. Drug supplied as a capsule taken orally.
  Other Names: Tecfidera; DMF; BG00012

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of BG00012 (dimethyl fumarate) administered in combination with interferon b (IFNß) or glatiramer acetate (GA) in participants with relapsing-remitting multiple sclerosis (RRMS).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of relapsing-remitting multiple sclerosis (RRMS) according to McDonald criteria #1-4 (Polman et al, 2005 [Appendix I]), and have a prior brain magnetic resonance imaging (MRI) demonstrating lesion (s) consistent with multiple sclerosis (MS) from any point in time.
* Must have an Expanded Disability Status Scale (EDSS) between 0.0 and 5.0, inclusive.
* Must be taking the same dose of a prescribed IFNβ (either Avonex, Betaseron, Rebif) or GA for at least 12 months consecutively at the time of enrollment and remain on this treatment for the duration of the study. Participants receiving Rebif must be prescribed 44 μg by subcutaneous injection three times per week.

Key Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS (as defined by Polman et al. 2005).
* Other chronic disease of the immune system, malignancies, acute urologic, or pulmonary disease.
* Pregnant or nursing women.
* Participation within 6 months prior to study enrollment in any other drug, biologic, or device study.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (16):
- United States (16):
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Danbury, Connecticut
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Golden Valley, Minnesota
  - Research Site, Teaneck, New Jersey
  - Research Site, Patchogue, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Cordova, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Background] Calkwood J, Vollmer T, Fox RJ, Zhang R, Novas M, Sheikh SI, Viglietta V. Safety and Tolerability of Delayed-Release Dimethyl Fumarate Administered with Interferon Beta or Glatiramer Acetate in Relapsing-Remitting Multiple Sclerosis. Int J MS Care. 2016 May-Jun;18(3):138-46. doi: 10.7224/1537-2073.2015-020. PMID 27252601

RESULTS

PARTICIPANT FLOW:
Groups:
- Monotherapy Period: Interferon Beta (IFNß): Participants taking a stable dose of one of the IFNß products for at least 12 months prior to the study remained on that product and dose throughout the study. The monotherapy period included the 8 weeks prior to the first dose of dimethyl fumarate.
- Monotherapy Period: Glatiramer Acetate (GA): Participants taking a stable dose of GA for at least 12 months prior to the study remained on that dose throughout the study. The monotherapy period included the 8 weeks prior to the first dose of dimethyl fumarate.
- Add-on Therapy Period: Dimethyl Fumarate Add-on to IFNß: BG00012 (dimethyl fumarate) was to be administered at 120 mg three times a day (TID) on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months) as an add-on to a stable dose of IFNß.
  Participants taking a stable dose of one of the IFNß products for at least 12 months prior to the study remained on that product and dose throughout the study.
- Add-on Therapy Period: Dimethyl Fumarate Add-on to GA: Dimethyl fumarate was to be administered at 120 mg TID on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
  Participants taking a stable dose of GA for at least 12 months prior to the study remained on that dose throughout the study.
Period: 2-Month Monotherapy Period
Arm/Group | Monotherapy Period: Interferon Beta (IFNß) | Monotherapy Period: Glatiramer Acetate (GA) | Add-on Therapy Period: Dimethyl Fumarate Add-on to IFNß | Add-on Therapy Period: Dimethyl Fumarate Add-on to GA
Started | 59 | 49 | 0 | 0
Completed | 57 | 47 | 0 | 0
Not Completed | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: 6-month Add-on Therapy Period
Arm/Group | Monotherapy Period: Interferon Beta (IFNß) | Monotherapy Period: Glatiramer Acetate (GA) | Add-on Therapy Period: Dimethyl Fumarate Add-on to IFNß | Add-on Therapy Period: Dimethyl Fumarate Add-on to GA
Started | 0 | 0 | 57 | 47
Completed BG00012 Combination Therapy | 0 | 0 | 45 | 38
Completed | 0 | 0 | 45 | 37
Not Completed | 0 | 0 | 12 | 10
Not completed — Adverse Event | 0 | 0 | 7 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Disease Activity | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: participants who took at least 1 capsule of BG00012 concurrently with the background therapy (combination therapy).
Groups:
- Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate): Participants taking a stable dose of one of the IFNß products for at least 12 months prior to the study remained on that product and dose throughout the study. BG00012 (dimethyl fumarate) was to be administered at 120 mg TID on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
- Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate): Participants taking a stable dose of GA for at least 12 months prior to the study remained on that dose throughout the study. BG00012 (dimethyl fumarate) was to be administered at 120 mg TID on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
- Total: Total of all reporting groups
Arm/Group | Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate) | Total
Number analyzed (Participants) | 57 | 47 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (7.58) | 40.7 (8.44) | 40.1 (7.96)
Age, Customized [Number; unit: participants]
  18 to 19 years | 1 | 0 | 1
  20 to 29 years | 5 | 3 | 8
  30 to 39 years | 18 | 22 | 40
  40 to 49 years | 27 | 15 | 42
  50 to 55 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 29 | 69
  Male | 17 | 18 | 35

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Summary of Adverse Events (AEs) Occurring Before BG00012 Dosing (Monotherapy Period)
Description: Percentage of participants with AEs, serious AEs (SAEs), and discontinuations due to AEs. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not related to the study drug. An SAE was any untoward medical occurrence that, at any dose: resulted in death; in the view of the Investigator, placed the participant at immediate risk of death (a life-threatening event); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; was any other medically important event that, in the opinion of the Investigator, jeopardized the participant or required intervention to prevent one of the other outcomes above. AEs were categorized as mild, moderate, or severe. All AEs occurring from enrollment to the day before BG00012 dosing are included.
Time Frame: from time of enrollment until day before first administration of BG00012 (Week -8 to Week 0)
Population: The Safety Population for the Monotherapy Period was defined as any participant who took at least 1 dose of background therapy.
Measure: Number; unit: percentage of participants
Groups:
- Monotherapy Period: IFNß: Participants taking a stable dose of one of the IFNß products for at least 12 months prior to the study remained on that product and dose throughout the study. The monotherapy period included the 8 weeks prior to the first dose of dimethyl fumarate.
- Monotherapy Period: GA: Participants taking a stable dose of GA for at least 12 months prior to the study remained on that dose throughout the study. The monotherapy period included the 8 weeks prior to the first dose of dimethyl fumarate.
Arm/Group | Monotherapy Period: IFNß | Monotherapy Period: GA
Number analyzed (Participants) | 59 | 49
percentage of participants
  Participants with an AE | 56 | 49
  Participants with a moderate or severe AE | 22 | 27
  Participants with a severe AE | 3 | 0
  Participants with an SAE | 0 | 0
  Participants withdrawing from study due to an AE | 0 | 0

2. Primary Outcome: Summary of Treatment-emergent Adverse Events (TEAEs) Occurring Post-BG00012 Dosing (Add-on Therapy Period)
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not related to the study drug. A serious adverse event (SAE) was any untoward medical occurrence that, at any dose: resulted in death; in the view of the Investigator, placed the participant at immediate risk of death (a life-threatening event); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; was any other medically important event that, in the opinion of the Investigator, jeopardized the participant or required intervention to prevent one of the other outcomes above. TEAE was defined as having an onset date that was on or after the start of study treatment (BG00012), or that worsened after the start of study treatment.
Time Frame: AEs were collected from enrollment until the final study visit (Week 26 +/-5 days).
Population: The Safety Population for the Combination Therapy Period was defined as any participant who took at least 1 capsule of BG00012 concurrently with the background therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate)
Number analyzed (Participants) | 57 | 47
percentage of participants
  Participants with a TEAE | 95 | 100
  Participants with a moderate or severe TEAE | 72 | 70
  Participants with a severe TEAE | 14 | 15
  Participants with a related TEAE | 74 | 87
  Participants with a serious TEAE | 4 | 2
  Participants discontinuing BG00012 due to a TEAE | 14 | 17
  Participants withdrawing from study due to a TEAE | 14 | 17

3. Primary Outcome: Potentially Clinically Significant Hematology Laboratory Abnormalities for Combination Therapy
Description: Percentage of participants with potentially clinically significant hematology laboratory abnormalities.
Time Frame: collected from the start of BG00012 administration through to Week 26 +/- 5 days
Population: Participants in the safety population with at least one post-baseline value. Safety Population for the Combination Therapy Period was defined as any participant who took at least 1 capsule of BG00012 concurrently with the background therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate)
Number analyzed (Participants) | 56 | 47
percentage of participants
  White Blood Cells (total) < 3.0*10^9/L | 9 | 2
  White Blood Cells (total) ≥ 16*10^9/L | 2 | 2
  Lymphocytes < 0.8*10^9/L | 32 | 6
  Lymphocytes < 0.5*10^9/L | 7 | 4
  Lymphocytes > 12*10^9/L | 0 | 0
  Neutrophils ≤ 1.0*10^9/L | 0 | 0
  Neutrophils < 1.5*10^9/L | 13 | 2
  Neutrophils ≥ 12*10^9/L | 2 | 4
  Red Blood Cells ≤ 3.3*10^12/L | 0 | 0
  Red Blood Cells ≥ 6.8*10^12/L | 0 | 0
  Hemoglobin g/L ≤ 100 | 0 | 0
  Platelet Count ≤ 100*10^9/L | 0 | 0
  Platelet Count ≥ 600*10^9/L | 0 | 0

4. Primary Outcome: Maximum Post-Baseline Values: Liver Enzymes for Combination Therapy
Description: Percentage of participants with post-baseline liver enzyme values above the upper limit of normal (ULN). Liver enzymes included alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), and bilirubin. Elevated ALT/AST (ALT/AST ≥ 3*ULN) concurrent with elevated total bilirubin was also evaluated.
Time Frame: collected from the start of BG00012 administration through to Week 26 +/- 5 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate)
Number analyzed (Participants) | 57 | 47
percentage of participants
  ALT ≤ 1*ULN | 47 | 47
  ALT > 1*ULN | 53 | 53
  ALT ≥ 3*ULN | 5 | 2
  ALT > 5*ULN | 2 | 0
  ALT > 10*ULN | 0 | 0
  ALT > 20*ULN | 0 | 0
  AST ≤ 1*ULN | 68 | 64
  AST > 1*ULN | 32 | 36
  AST ≥ 3*ULN | 2 | 0
  AST > 5*ULN | 0 | 0
  AST > 10*ULN | 0 | 0
  AST > 20*ULN | 0 | 0
  GGT ≤ 1*ULN | 72 | 85
  GGT > 1*ULN | 28 | 15
  GGT ≥ 3*ULN | 4 | 0
  GGT > 5*ULN | 2 | 0
  GGT > 10*ULN | 0 | 0
  GGT > 20*ULN | 0 | 0
  Total Bilirubin ≤ 1*ULN | 98 | 94
  Total Bilirubin > 1*ULN | 2 | 6
  Total Bilirubin > 1.5*ULN | 0 | 4
  Total Bilirubin > 2*ULN | 0 | 2
  ALT/AST ≥ 3*ULN + Total Bilirubin > 1.5*ULN | 0 | 0
  ALT/AST ≥ 3*ULN + Total Bilirubin > 2*ULN | 0 | 0

5. Primary Outcome: Worst Post-Baseline Values for Selected Urinalysis Parameters That Require Further Evaluation for Combination Therapy
Description: Percentage of participants with post-baseline values for selected urinalysis parameters requiring further evaluation. For urine microscopy, results were categorized for male and female participants. For males, normal/negative was considered 0 to 3 red blood cells/high-power field (rbc/hpf), and positive was categorized in the following stages: 4 to 10, 11 to 20, 21 to 149, and ≥ 150 rbc/hpf. For females, normal/negative was considered 0 to 8 rbc/hpf, and positive was categorized in the following stages: 9 to 20, 21 to 30, 31 to 149, and ≥ 150 rbc/hpf.
Time Frame: collected from the start of BG00012 administration through to Week 26 +/- 5 days
Population: The Safety Population for the Combination Therapy Period was defined as any participant who took at least 1 capsule of BG00012 concurrently with the background therapy; n=participants in the safety population with at least 1 post-baseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate)
Number analyzed (Participants) | 57 | 47
percentage of participants
  Urine blood: normal/negative; n=57, 47 | 75 | 64
  Urine blood: trace; n=57, 47 | 7 | 9
  Urine blood: 1+; n=57, 47 | 5 | 15
  Urine blood: 2+; n=57, 47 | 7 | 11
  Urine blood: 3+; n=57, 47 | 5 | 2
  Urine protein: normal/negative; n=57, 47 | 39 | 38
  Urine protein: trace; n=57, 47 | 35 | 45
  Urine protein: 1+; n=57, 47 | 26 | 15
  Urine protein: 2+; n=57, 47 | 0 | 2
  Urine protein: 3+; n=57, 47 | 0 | 0
  Urine protein: 4+; n=57, 47 | 0 | 0
  Urine glucose: normal/negative; n=57, 47 | 93 | 94
  Urine glucose: trace; n=57, 47 | 2 | 0
  Urine glucose: 1+; n=57, 47 | 2 | 2
  Urine glucose: 2+; n=57, 47 | 0 | 4
  Urine glucose: 3+; n=57, 47 | 2 | 0
  Urine glucose: 4+; n=57, 47 | 2 | 0
  Urine ketone: normal/negative; n=57, 47 | 47 | 57
  Urine ketone: trace; n=57, 47 | 9 | 11
  Urine ketone: 1+; n=57, 47 | 26 | 28
  Urine ketone: 2+; n=57, 47 | 11 | 4
  Urine ketone: 3+; n=57, 47 | 4 | 0
  Urine ketone: 4+; n=57, 47 | 4 | 0
  Urine microscopy (male): 0-3 rbc/hpf; n=9, 16 | 100 | 75
  Urine microscopy (male): 4-10 rbc/hpf; n=9, 16 | 0 | 6
  Urine microscopy (male): 11-20 rbc/hpf; n=9, 16 | 0 | 13
  Urine microscopy (male): 21-149 rbc/hpf; n=9, 16 | 0 | 6
  Urine microscopy (male): ≥ 150 rbc/hpf; n=9, 16 | 0 | 0
  Urine microscopy (female): 0-8 rbc/hpf; n=25, 28 | 76 | 86
  Urine microscopy (female): 9-20 rbc/hpf; n=25, 28 | 8 | 4
  Urine microscopy (female): 21-30 rbc/hpf; n=25, 28 | 4 | 0
  Urine microscopy (female): 31-149 rbc/hpf;n=25, 28 | 0 | 7
  Urine microscopy (female): ≥150 rbc/hpf; n=25, 28 | 12 | 4

6. Other Pre Specified Outcome: Average Number of Gadolinium (Gd)-Enhancing Lesions: Week -8, -4, 0 Average Versus Week 16, 20, 24 Average
Description: The average is calculated as (total number of lesions in non-missing scans / number of non-missing magnetic resonance imaging [MRI] scans).
Time Frame: Week -8 through Week 24
Population: Gd cohort: BG00012-dosed participants with at least 1 Gd-enhancing lesion in any 1 of the 3 scans (Weeks -8, -4, or 0) during the Monotherapy Period.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate)
Number analyzed (Participants) | 16 | 18
lesions
  Average number of lesions from Weeks -8, -4, 0 | 1.06 (1.011) | 1.72 (1.098)
  Average number of lesions from Weeks 16, 20, 24 | 0.17 (0.243) | 0.83 (2.115)
  Change from average of Weeks -8, -4, 0 | -0.90 (0.902) | -0.89 (2.264)
Statistical Analysis 1: Comparison: Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate); Change from average of Weeks -8, -4, and 0 to average of Weeks 16, 20, 24 MRI scans; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test; Median Difference (Final Values) = -0.92, 95% CI 2-sided [-1.17 to -0.33] — based on Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate); Change from average of Weeks -8, -4, and 0 to average of Weeks 16, 20, 24 MRI scans; Test type: Superiority or Other; p = 0.0124, Wilcoxon signed rank test; Median Difference (Final Values) = -1.17, 95% CI 2-sided [-1.83 to -0.33] — based on Hodges-Lehmann estimate

7. Other Pre Specified Outcome: Average Number of New Gd-Enhancing Lesions: Weeks -4, 0 Average Versus Weeks 20, 24 Average
Description: The average is calculated as (total number of lesions in non-missing scans / number of non-missing MRI scans).
Time Frame: Week -4 through Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate)
Number analyzed (Participants) | 16 | 17
lesions
  Average number of lesions from Weeks -4, 0 | 0.91 (0.953) | 0.79 (0.985)
  Average number of lesions from Weeks 20, 24 | 0.06 (0.171) | 0.18 (0.303)
  Change from average of Weeks -4, 0 | -0.84 (0.978) | -0.62 (1.054)
Statistical Analysis 1: Comparison: Interferon Beta (IFNß) and BG00012 (Dimethyl Fumarate); Change from average of Weeks -4, and 0 to average of Weeks 20, 24 MRI scans; Test type: Superiority or Other; p = 0.0010, Wilcoxon signed rank test; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-1.50 to -0.25] — based on Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate); Change from average of Weeks -4, and 0 to average of Weeks 20, 24 MRI scans; Test type: Superiority or Other; p = 0.0339, Wilcoxon signed rank test; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-1.25 to 0.00] — based on Hodges-Lehmann estimate

8. Other Pre Specified Outcome: Number of New or Newly Enlarging T2 Lesions
Description: The number of new T2 lesions divided by the number of months since the reference visit during the Monotherapy Period and the Add-On Therapy Period.
Time Frame: Week -8 to Week 24
Population: Number of participants in the Gd cohort with analyzable data in both Monotherapy and Add-on Therapy Periods. Gd cohort: BG00012-dosed participants with at least 1 Gd-enhancing lesion in any 1 of the 3 scans (Weeks -8, -4, or 0) during the Monotherapy Period.
Measure: Mean (Standard Deviation); unit: lesions per month
Groups:
- Interferon Beta 1a (IFNß) and BG00012 (Dimethyl Fumarate): Participants taking a stable dose of one of the IFNß products for at least 12 months prior to the study remained on that product and dose throughout the study. BG00012 (dimethyl fumarate) was to be administered at 120 mg TID on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
Arm/Group | Interferon Beta 1a (IFNß) and BG00012 (Dimethyl Fumarate) | Glatiramer Acetate (GA) and BG00012 (Dimethyl Fumarate)
Number analyzed (Participants) | 15 | 18
lesions per month
  New lesions in the Monotherapy Period | 1.23 (1.498) | 0.89 (1.243)
  New lesions in the Add-on Therapy Period | 0.67 (1.257) | 0.25 (0.293)

ADVERSE EVENTS:
Time Frame: AEs for the Monotherapy Period collected from enrollment until prior to administration of BG00012. TEAEs for the Add-on Therapy Period collected from start of BG00012 until the final study visit (Week 26 +/-5 days).
Description: AEs for the Monotherapy Period were summarized for all enrolled participants and were included for completeness only. No direct comparisons were made between the 2-month Monotherapy and the 6-month Add-on Therapy Periods due to the difference in the length of observation between these 2 periods.
Groups:
- Monotherapy Period: IFNß: A stable dose of one of the IFNß products for up to 8 weeks (until the first dose of BG00012).
- Monotherapy Period: GA: A stable dose of GA for up to 8 weeks (until the first dose of BG00012).
- Add-on Therapy Period: IFNß and BG00012: Participants taking a stable dose of one of the IFNß products for at least 12 months prior to the study remained on that product and dose throughout the study. BG00012 (dimethyl fumarate) was to be administered at 120 mg TID on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
- Add-on Therapy Period: GA and BG00012: Participants taking a stable dose of GA for at least 12 months prior to the study remained on that dose throughout the study. BG00012 (dimethyl fumarate) was to be administered at 120 mg TID on Days 1-7, and 240 mg TID on Day 8 until the end of treatment (approximately 6 months).
Arm/Group | Monotherapy Period: IFNß | Monotherapy Period: GA | Add-on Therapy Period: IFNß and BG00012 | Add-on Therapy Period: GA and BG00012
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/49 | 2/57 | 1/47
Other Adverse Events (participants affected / at risk) | 13/59 | 7/49 | 53/57 | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Period: IFNß (N=59) | Monotherapy Period: GA (N=49) | Add-on Therapy Period: IFNß and BG00012 (N=57) | Add-on Therapy Period: GA and BG00012 (N=47)
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Period: IFNß (N=59) | Monotherapy Period: GA (N=49) | Add-on Therapy Period: IFNß and BG00012 (N=57) | Add-on Therapy Period: GA and BG00012 (N=47)
Urinary Tract Infection (Infections and infestations) | 3 | 4 | 2 | 7
Nasopharyngitis (Infections and infestations) | 3 | 1 | 8 | 7
Multiple Sclerosis Relapse (Nervous system disorders) | 8 | 2 | 10 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 7 | 6
Sinusitis (Infections and infestations) | 0 | 0 | 4 | 6
Ear Infection (Infections and infestations) | 0 | 0 | 3 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 0 | 0 | 9 | 7
Dizziness (Nervous system disorders) | 0 | 0 | 8 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 4 | 3
Balance Disorder (Nervous system disorders) | 0 | 0 | 4 | 2
Migraine (Nervous system disorders) | 0 | 0 | 2 | 4
Paraesthesia (Nervous system disorders) | 0 | 0 | 3 | 1
Decreased Vibratory Sense (Nervous system disorders) | 0 | 0 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 3 | 1
Flushing (Vascular disorders) | 0 | 0 | 24 | 25
Hot Flush (Vascular disorders) | 0 | 0 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 18 | 7
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 12 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 11 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 8 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 7 | 4
Flatulence (Gastrointestinal disorders) | 0 | 0 | 4 | 6
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 4 | 5
Constipation (Gastrointestinal disorders) | 0 | 0 | 5 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Fatigue (General disorders) | 0 | 0 | 8 | 4
Pyrexia (General disorders) | 0 | 0 | 5 | 1
Pain (General disorders) | 0 | 0 | 3 | 2
Chills (General disorders) | 0 | 0 | 4 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 6 | 7
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 4 | 4
Gamma-glutamyltransferase Increased (Investigations) | 0 | 0 | 2 | 3
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 5 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 3 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.